CLINICAL TRIAL: NCT03183427
Title: Corpus Callosum Size in Patients With Pineal Cyst
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Military University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Martin Majovsky, MD, Senior physician, Military University Hospital, Prague
Other Study IDs: 108/11-28/2017
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Pineal Gland Disorder; Corpus Callosum Atrophy; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of patients with pineal cyst: Group of patients with pineal cyst
  Interventions: Diagnostic Test: MR of the brain
- Control group: Group of subjects without pineal cyst
  Interventions: Diagnostic Test: MR of the brain

INTERVENTIONS:
Diagnostic Test: MR of the brain — MR of the brain without gadolinium, incl. T2-weighted image

SUMMARY:
This study aims to determine size of corpus callosum on midsagittal MR scan in patients with a pineal cyst and to compare it with the control group without a pineal cyst.

DETAILED DESCRIPTION:
A pineal cyst (PC) is a benign affection of the pineal gland, its prevalence in population reaches 1-2 %. Etiopathogenesis of PC is unknown, several hypotheses have been proposed. One of the hypothesis consider perinatal hypoxia as a causative factor for a development of PC in later life. Ozmen et al. showed significantly higher prevalence of PC in patients with cerebral palsy (p<0.001). Bregant et al. studied presence of PC in patients that suffered from a mild to moderate perinatal hypoxia. Prevalence of PC reached 36 % in these patients and presence of PC was associated with a atrophy of the corpus callosum (p<0.005). The atrophy of the corpus callosum is considered to be a sign of a periventricular leukomalacia, i.e. an ischemic insult in a perinatal period.

In the present study, we are going to compare an area of corpus callosum on a midsagittal magnetic resonance T2-weighted scan in the group of patients with PC and in the control group without PC. The goal of the study is to determine if there is a relationship between atrophy of the corpus callosum and PC. Such finding would support abovementioned theory of etiopathogenesis of PC.

ELIGIBILITY:
Inclusion Criteria:

* 3T MR examination of the brain including T2 sagittal scans

Exclusion Criteria:

* other intracranial pathology discovered on the MR
* other known neurological disease (e.g. multiple sclerosis, stroke, tumor, etc.)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * study group: consecutive patients with pineal cyst that were examined in our institution between 2000-2017
  * control group: matched healthy subjects without pineal cyst
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
size of corpus callosum | time of the MR examination
  size of corpus callosum in mm2 measured on the midsagittal T2-weighted MR scan

IPD SHARING:
Plan to Share IPD: No